CLINICAL TRIAL: NCT03381209
Title: The Effect of Sugammadex Given Based on Ideal, Actual or Adjusted Body Weights on Reversal of Neuromuscular Blockade in Morbidly Obese Patients Undergoing Laparoscopic Bariatric Surgery
Brief Title: The Effect of Sugammadex Given Based on Ideal, Actual or Adjusted Body Weight on Reversal of Rocuronium.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Walid Nofal, Lecturer of Anesthesiology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FMASU R 39/2017
Record Dates: First submitted 2017-12-17; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Muscle Relaxation
Keywords: Sugammadex; morbidly obese patients; bariatric surgery; neuromuscular blockade
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Sugammadex given in a dose of 2mg/kg based on ideal body weight
  Interventions: Drug: Sugammadex
- Group B (Experimental): Sugammadex given in a dose of 2mg/kg based on adjusted body weight
  Interventions: Drug: Sugammadex
- Group C (Experimental): Sugammadex given in a dose of 2mg/kg based on actual body weight
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — sugammadex given based on 3 measurements of body weights
  Other Names: bridion

SUMMARY:
The aim of this study is compare the reversal of rocuronium induced neuromuscular blockade in morbidly obese patients using three doses of sugammadex; based on ideal body weight, adjusted body weight, and actual body weight.

DETAILED DESCRIPTION:
The aim of this study is compare the reversal of rocuronium induced neuromuscular blockade in morbidly obese patients using three doses of sugammadex; based on ideal body weight, adjusted body weight, and actual body weight. Reversal Time: time from administration of Sugammadex to train of four (TOF) ratio ≥ 0.9 will be used as primary outcome.

Time need for extubation (time from administration of sugammadex to extubation), and duration of stay in post anesthesia care unit (PACU), will be used as secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years and under 45 years,
* body mass index ≥ 40 kg/m2, with indication of bariatric surgery

Exclusion Criteria:

* Patients with comorbid including: neuromuscular disease, renal impairment, and patients with difficult airway were excluded from this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Reversal Time | 5 minutes after sugammadex administration
  Reversal Time: time from administration of Sugammadex to train of four (TOF) ratio ≥ 0.9 will be used as primary outcome.

SECONDARY OUTCOMES:
duration of stay in PACU | 60 minutes after admission to the PACU
  period of stay in the PACU
Time need for Extubation | 10 minutes after sugammadex administration
  time from administration of sugammadex to extubation

CONTACTS AND LOCATIONS:
Overall Officials: Walid Nofal, MD, Principal Investigator — Anesthesiology department, Faculty of Medicine, Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No